CLINICAL TRIAL: NCT01247883
Title: A Two Period, 2 Sequence Crossover To Establish The Relative Bioavailability Of A Single Pf-04634817 Tablet Dose Compared With A Solution In Healthy Volunteers
Brief Title: A Comparison Of A Single PF-04634817 Tablet Dose Compared With A Solution In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1261005
Record Dates: First submitted 2010-10-20; First posted 2010-11-24 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Phase 1; relative bioavailability; healthy volunteers; pharmacokinetics; solution; tablet
MeSH Terms: interventions — PF-04634817

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single dose PF-04634817 tablet (Active Comparator): subjects receive a single dose of PF-04634817 as a tablet
  Interventions: Drug: PF-04634817
- single dose PF-04634817 solution (Active Comparator): subjects receive a single dose of PF-04634817 as a solution
  Interventions: Drug: PF-04634817

INTERVENTIONS:
Drug: PF-04634817 — single dose, 20mg, tablet
  Arms: single dose PF-04634817 tablet
Drug: PF-04634817 — single dose, 20mg, solution
  Arms: single dose PF-04634817 solution

SUMMARY:
This study investigates the safety, tolerability and pharmacokinetics of PF-04634817 when respectively given orally as a single tablet dose and a single dose of a solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history and full physical examination.)
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication;
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day;
* Nursing females;
* Females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
adverse events | 4 days
Plasma Pharmacokinetics for both tablet and solution dosage forms. | 4 days
The relative bioavailability (Frel) of PF-04634817 when administered as a tablet compared with a solution. | 4 days
lab measurements | 4 days
vitals/ECG parameters | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261005&StudyName=A%20comparison%20Of%20A%20single%20PF-04634817%20Tablet%20Dose%20Compared%20With%20A%20Solution%20In%20Healthy%20Volunteers%20